## "Graviditetskomplikationer - en probiotisk interventionsstudie"

## Patientens samtycke till att delta i studien:

Jag har muntligen informerats om studien och tagit del av den skriftliga informationen. Jag är medveten om att mitt deltagande i studien är frivilligt, och att jag när som helst och utan närmare förklaring kan avbryta mitt deltagande utan att det påverkar mitt omhändertagande. Jag har haft möjlighet att ställa frågor om studien och fått dem besvarade.

Jag har informerats om och samtycker till att berörd forskningspersonal studerar mina och mitt blivande barns medicinska journaler.

Jag har informerats om de prover som skall tas och att jag när som helst och utan närmare förklaring kan begära att dessa prover förstörs. Jag har informerats om att proverna hanteras enligt biobankslagen.

Jag har informerats om risker och fördelar med studien. Jag har förstått den information jag fått och jag samtycker till att delta i studien.

| Underskrift av patient: | |
|---|---|
| Namnförtydligande av patient: | |
| Datum: | |
| A | |
| Ansvarig prövares försäkran: | |
| Jag intygar att jag lämnat fullständig information om den pågående studien till ovanstående patie Jag har gått igenom och förklarat studiens syfte för patienten. Patienten har haft möjlighet att stä frågor och fått dem besvarade. Patienten har fått en kopia på den skriftliga patientinformationen kopia på samtyckesformuläret kommer att finnas i patientens journal. | älla |
| Underskrift av ansvarig prövare: | |
| Namnförtydligande av ansvarig prövare: | |
| Datum: | |